CLINICAL TRIAL: NCT05204095
Title: Intelligent Cataract Screening With Portable Slit-lamp
Acronym: AI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: SLCS-2022
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Catarct Screening; Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Referral group: The patients with severe cataracts in this group need a referral to a higher-level hospital for further treatment.
  Interventions: Device: Portable slit-lamp photography
- Observation group: The patients with mild cataracts or transparent lenses in this group do not need a referral to a higher-level hospital for further treatment and keep regular examinations.
  Interventions: Device: Portable slit-lamp photography

INTERVENTIONS:
Device: Portable slit-lamp photography — The enrolled patients will undergo portable slit-lamp photography with and without mydriasis and receive traditional slit-lamp photography for comparison.

SUMMARY:
Based on the portable slit-lamp connected to the smartphone, the artificial intelligence machine learning algorithm is used to establish a cataract screening model by prospectively collecting the anterior segment photographic data, and a portable slit lamp intelligent screening referral model based on the smartphone connection is also established.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 100 years old

Exclusion Criteria:

* (1) History of eye disease except for age-related cataracts (2) History of eye trauma or eye surgery (3) Unable to cooperate with ophthalmology and general examination (4) Individuals with incomplete information (5) Unwilling to participate in this study

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The prospective population aged 0 to 100 with or without senile cataracts and received ocular examination.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of referral | Baseline
  The accuracy of referral of AI model will be calculated with the decisions based on the portable slit-lamp images with reference to the ground truth.

SECONDARY OUTCOMES:
The accuracy of cataract diagnosis | Baseline
  The accuracy of cataract diagnosis of AI model will be calculated with the decisions based on the portable slit-lamp images with reference to the ground truth.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China